CLINICAL TRIAL: NCT04427033
Title: The BCI 602 BONEBRIDGE Post-Market Clinical Follow-up Study
Status: Completed | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019BB005
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed; Hearing Loss, Unilateral; Hearing Loss, Bilateral; Hearing Loss, Sensorineural
Keywords: Bonebridge system; BCI 601; BCI 602; bone conduction; bone conduction implant
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Unilateral; Hearing Loss, Bilateral; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- CHL & MHL (18 years and older): CHL= conductive hearing loss, MHL= mixed hearing loss
  Interventions: Device: Bone Conduction Implant
- CHL & MHL (5 to 17 years)
  Interventions: Device: Bone Conduction Implant
- SSD (5 years and older): SSD= single sided deafness
  Interventions: Device: Bone Conduction Implant

INTERVENTIONS:
Device: Bone Conduction Implant — Bonebridge system BCI 602

SUMMARY:
The Bonebridge system using the BCI 601 is marketed since 2012. Previous prospective, multi-center, non-randomized studies on the BCI 601 Bonebridge performed in adult and paediatric populations have shown a significant improvement in terms of aided sound field (SF) thresholds, word recognition scores (WRS), speech reception thresholds (SRT) and subjective device satisfaction. Safety was established by stable residual hearing and low complication rates. The Bonebridge, implanted in over 600 clinics worldwide, is the world's first active transcutaneous bone conduction implant (BCI) system.

This study now focuses on the further developed BCI 602 (marketed since 2019) that has the same indication criteria and performance characteristics.

The aim of this post-market clinical follow-up (PMCF) study is to provide clinical data for the long-term performance and safety when implanted with the Bonebridge BCI 602 .

ELIGIBILITY:
Inclusion Criteria:

* Geographically and physically able to return to the investigational site for scheduled evaluations and follow-up appointments
* Fluent in the language used in the investigational site and used for evaluation
* Signed and dated informed consent before the start of any study-specific procedure and collection of any retrospective data.
* Subjects meet the indication criteria according to the instructions for use (IFU):

  * Subject 5 years of age and older
  * The physician must fully assess the potential risks and benefits for the patient and his/her realistic expectations with the device prior to the decision to implant the BCI 602. The physician must exercise medical judgement and consider the patient's complete medical history.
  * Bonebridge candidates suffer from either
  * • conductive or mixed hearing loss as indicated by audiometric testing with bone conduction thresholds better than or equal to 45 dB HL at 0.5, 1.0, 2.0 and 3.0 kHz.
  * • single-sided sensorineural deafness, that is severe-to-profound sensorineural hearing loss in one ear while the other ear has normal hearing (air conduction (AC) should be better than or equal to 20 dB HL measured at 0.5, 1.0, 2.0 and 3.0 kHz).

Exclusion Criteria:

* A subject whose hearing loss has demonstrated an improving and decreasing fluctuation over a two-year period of >15 dB HL in either direction
* Severe, chronic, non-revisable diseases or disorders (vestibular disorder, cancer etc.)
* A subject with any psychological (anxiety, depression, hallucinations etc.), emotional (schizophrenia, mania, melancholia etc.) or from that originating physical disorder that would interfere with the ability to perform on test procedures
* Simultaneous participation in another clinical trial (on device or on drug) which would interfere with the results of the study.
* Any active ear infection
* Subjects who meet any of the contraindications in the IFU:

  * Evidence that hearing loss is of retrocochlear or central origin (ipsilateral CHL /MHL; contralateral SSD)
  * Skin or scalp conditions that may preclude attachment of the Audio Processor (AP) or that may interfere with the use of the AP
  * Skull size or abnormality would preclude appropriate placement of the BCI 602 implant
  * Intolerant to the materials in the BCI 602 implant.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will only enrol subjects who represent the target population and meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Sound Field audiometry | 12 months post-operative
  Investigate if the PTA4 sound field thresholds (SF) improve with the BCI 602 (aided) at 12 months post-operative compared to the unaided test situation.
  (PTA4 = average of audiometric test frequencies 0.5, 1.0, 2.0, 4.0 kHz)

SECONDARY OUTCOMES:
Word Recognition Score (CHL/MHL) | 12 months post-operative
  Investigate if speech intelligibility improves with the BCI 602 (aided) at 12 months post-operative compared to the unaided test situation in the following speech intelligibility test.
  Word Recognition Score (WRS): S0°, WRS correct @ 65 dB SPL Signal
  Monosyllabic (MS) word lists are presented from the front (0°) at 65 dB SPL (45 dB HL) and the percent correct score [%] (0 % to 100 %) is recorded.
  (SPL= Sound Pressure Level; Score: 0% to 100% words understood )
Speech Reception Threshold in quiet (CHL/MHL) | 12 months post-operative
  Investigate if speech intelligibility improves with the BCI 602 (aided) in CHL/MHL at 12 months post-operative compared to the unaided test situation in the following speech intelligibility test.
  Speech Reception Threshold in quiet (SRT) : S0°, SRT for 50% correct
Speech Reception Threshold in noise (CHL/MHL) | 12 months post-operative
  Investigate if speech intelligibility improves with the BCI 602 (aided) in CHL/MHL at 12 months post-operative compared to the unaided test situation in the following speech intelligibility test.
  Speech Reception Threshold in noise (SNR): S0° N0°, SNR for 50% correct @ 65 dB SPL Noise
Speech Reception Threshold in noise (SSD) Sssd Nnh | 12 months post-operative
  Investigate if speech intelligibility improves with the BCI 602 (aided) in SSD at 12 months post-operative compared to the unaided test situation in the following speech intelligibility tests.
  Sssd Nnh, SNR for 50% correct @ 65 dB SPL Noise
  (S= Signal; N= Noise; ssd = single sided deaf ear; nh = normal hearing ear)
Speech Reception Threshold in noise (SSD) S0° Nnh | 12 months post-operative
  Investigate if speech intelligibility improves with the BCI 602 (aided) in SSD at 12 months post-operative compared to the unaided test situation in the following speech intelligibility tests.
  S0° Nnh, SNR for 50% correct @ 65 dB SPL Noise
Residual hearing | 12 months post-operative
  Investigate whether residual hearing by means of bone conduction (BC) PTA4 thresholds of subjects implanted with the BCI 602 remains stable 12 months post-operative compared to the pre operative test situation.
Adverse Events | 12 months post-operative
  Monitor the long-term safety of subjects implanted with the BCI 602 by collecting and reviewing adverse events (AEs).
Surgical Questionnaires | 12 months post-operative
  Monitor the long-term safety of subjects implanted with the BCI 602 by administering a surgical evaluation questionnaire to the surgeon.
Speech Spatial Qualities questionnaire | 12 months post-operative
  Investigate the Quality of Life with the SSQ questionnaire of subjects implanted with the BCI 602 12 months post-operative.
  (SSQ = Speech Spatial Qualities)
Assessment Quality of Life questionnaire | 12 months post-operative
  Investigate the Quality of Life with the AQoL questionnaire of subjects implanted with the BCI 602 12 months post-operative.
  (AQoL= Assessment Quality of Life)

CONTACTS AND LOCATIONS:
Overall Officials: Assen Koitschev, Prof. Dr., Principal Investigator — Klinikum Stuttgart - Olgahospital and Eberhard-Karls-Universität Tübingen
Locations (8):
- Austria (4):
  - Universitätsklinik Innsbruck für Hals-, Nasen- und Ohrenheilkunde, Innsbruck
  - Universitätsklinikum St. Pölten - Lilienfeld, Hals-Nasen-Ohren-Abteilung, Sankt Pölten
  - Allgemeines Krankenhaus der Stadt Wien, Universitätsklinik für Hals-, Nasen- und Ohrenkrankheiten, Vienna
  - Klinikum Wels-Grieskirchen, Abteilung für Hals-, Nasen-, Ohrenkrankheiten, Wels
- Germany (3):
  - Universitätsklinik und Poliklinik für Hals-Nasen-Ohren-Heilkunde, Kopf- und Hals-Chirurgie, Halle
  - Klinik u. Poliklinik f. HNO-Heilkunde, Hanover
  - Klinikum Stuttgart - Olgahospital, Klinik für HNO-Krankheiten, Plastische Operationen, Stuttgart
- Regional Auditory Implant Centre, Beech Hall Centre, Belfast HSC Trust, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sprinzl G, Lenarz T, Ernst A, Hagen R, Wolf-Magele A, Mojallal H, Todt I, Mlynski R, Wolframm MD. First European multicenter results with a new transcutaneous bone conduction hearing implant system: short-term safety and efficacy. Otol Neurotol. 2013 Aug;34(6):1076-83. doi: 10.1097/MAO.0b013e31828bb541. PMID 23714710
- [Background] Baumgartner WD, Hamzavi JS, Boheim K, Wolf-Magele A, Schlogel M, Riechelmann H, Zorowka P, Koci V, Keck T, Potzinger P, Sprinzl G. A New Transcutaneous Bone Conduction Hearing Implant: Short-term Safety and Efficacy in Children. Otol Neurotol. 2016 Jul;37(6):713-20. doi: 10.1097/MAO.0000000000001038. PMID 27153327
- [Background] Sprinzl G, Toner J, Koitschev A, Berger N, Keintzel T, Rasse T, Baumgartner WD, Honeder C, Magele A, Plontke S, Gotze G, Schmutzhard J, Zelger P, Corkill S, Lenarz T, Salcher R. Multicentric study on surgical information and early safety and performance results with the Bonebridge BCI 602: an active transcutaneous bone conduction hearing implant. Eur Arch Otorhinolaryngol. 2023 Apr;280(4):1565-1579. doi: 10.1007/s00405-022-07792-y. Epub 2023 Jan 10. PMID 36625869